CLINICAL TRIAL: NCT03475745
Title: The Usage of High-resolution Magnetic Resonance Imaging in Patients With Post-stroke Aphasia for Predicting the Outcome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: HRMRI- aphasia
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2017-11

CONDITIONS: Aphasia
Keywords: resting-state; DTI; aphasia; stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aphasia: Post stroke aphasia patients without any additional interventions for research purposes.
- Control: Healthy controls

SUMMARY:
Combined analysis of functional and structural language network changes may be a good model for predicting language outcome.

DETAILED DESCRIPTION:
Background & objectives:

Language impairment after aphasic stroke is both common and debilitating. However the mechanisms of language recovery after aphasic stroke is not fully understood. Investigators plan to detect the changes of functional and structural language networks after aphasic stroke by high-resolution MRI.Then Combined analyse functional and structural language network changes, establishing a prediction model for language outcome.

Methods:

The proposed study is a observational trial that will include 50 patients diagnosed with post stroke aphasia from the neurology clinics at The First Affiliated Hospital, Zhejiang University. Aphasia battery of Chinese(ABC) and functional magnetic resonance imaging (MRI) will be performed at acute(~2weeks),subacute(3 months) and chronic phase(6months). Only routine drug therapy will be used.

Relevance:

Currently there is little known about the recovery mechanisms of post-stroke aphasia.The proposed study intends to analyse functional and structural language network changes by high resolution MRI, which may reveal the potential recovery mechanism underlying post stroke aphasia..

ELIGIBILITY:
Inclusion Criteria:

* Healthy right-handed native Chinese speakers with more than 6-year education are recruited as healthy controls.

Exclusion Criteria:

* Not right-handed;
* Any use of psychoactive drugs;
* Less than 6-year education;
* Not suitable for MRI scan.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In-patients from Neurology departments of the First Affiliated Hospital, Zhejiang University
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Resting state functional connectivity changes | 3 months
  The study uses resting state functional MRI(rs-fMRI) to measure changes of functional connectivity across regions after a spontaneous recovery.

SECONDARY OUTCOMES:
Aphasia Battery of Chinese, ABC | 3 months
  ABC, the Chinese standardized adaptation of the Western Aphasia Battery, indicates the patient's ability of spontaneous speech, auditory comprehension, repetition, naming, reading, writing.
White matter Integrity | 3 months
  The study uses Diffusion tensor imaging and tracking (DTI) to measure changes of the Integrity of white matter after a spontaneous recovery.
Brain response change | 3 months
  The study uses task functional MRI (fMRI) to measure the brain response changes during the task after a spontaneous recovery.
Resting state functional connectivity changes | 6 months
  The study uses resting state functional MRI(rs-fMRI) to measure changes of functional connectivity across regions after a spontaneous recovery.
Aphasia Battery of Chinese, ABC | 6 months
  ABC, the Chinese standardized adaptation of the Western Aphasia Battery, indicates the patient's ability of spontaneous speech, auditory comprehension, repetition, naming, reading,
White matter Integrity | 6 months
  The study uses Diffusion tensor imaging and tracking (DTI) to measure changes of the Integrity of white matter after a spontaneous recovery.
Brain response change | 6 months
  The study uses task functional MRI (fMRI) to measure the brain response changes during the task after a spontaneous recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Ph.D, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No